CLINICAL TRIAL: NCT03355807
Title: Use of MgSO4 Reduced Opioid Consumption for Pain After Sleeve Gastrectomy Operations: A Prospective Randomized Clinical Trial
Brief Title: Use of MgSO4 for Pain After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, nurcan kizilcik, Assist. Prof. Dr., Yeditepe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: obesity (magnesium)
Record Dates: First submitted 2017-09-28; First posted 2017-11-28 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Therapeutic Opioid Induced Constipation (Disorder)
Keywords: sleeve gastrectomy; magnesium sulfate; postoperative pain; bariatric surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium

STUDY DESIGN:
Intervention Model Description: The patients undergoing sleeve gastrectomy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Patient, investigator and anesthesiologist who was blinded to the assignment of the patients recorded levels of sedation, pain, cumulative morphine consumption, and hemodynamic variables
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group MgSO4 (Experimental): The magnesium group (group Mg, n _ 40) received an additional infusion of MgSO4 (30 mg/kg by bolus and 10 mg/kg/h by infusion for 24 hours)
  Interventions: Drug: Magnesium
- Group Control (No Intervention): the control group (group C, n _ 40) received the same amount of IV saline

INTERVENTIONS:
Drug: Magnesium — The magnesium group (group Mg, n _ 40) received an additional infusion of MgSO4
  Arms: Group MgSO4

SUMMARY:
The purpose of this study was to investigate the effect of magnesium sulfate on pain management for pain after sleeve gastrectomy operation

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of magnesium sulfate on pain management for pain after sleeve gastrectomy operation.

Design: A prospective, randomized, controlled clinical study.

Setting: University hospital.

Participants: Eighty patients undergoing sleeve gastrectomy.

Measurements and Main Results: Visual analog scale for pain score, sedation score, mean arterial pressure, heart rate, and valid and invalid analgesic demand will record. Serum magnesium levels will determined at preoperative evaluation, postanesthesia care unit admission and at 24 hours. Side effects will also record.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 year old individuals who underwent laparoscopic sleeve gastrectomy.

Exclusion Criteria:

* One or more of the following: cardio - vascular and respiratory diseases, drug and/or alcohol abuse, use of daily an algesia 24 hours before the surgery, renal failure, and liver dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Item pain intensity measure assessed by using VAS scores | 1 day
  Pain was assessed by using VAS scores (0: no pain and 10: worst pain) imaginable recorded at 0, 1, 2, 4, 6, 24, and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: nurcan kizilcik, MD, Principal Investigator — yeditepe universityiversity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvarez A, Singh PM, Sinha AC. Postoperative analgesia in morbid obesity. Obes Surg. 2014 Apr;24(4):652-9. doi: 10.1007/s11695-014-1185-2. PMID 24431032
- See also: bariatric surgery and anesthesia — http://bariatrictimes.com